CLINICAL TRIAL: NCT04712214
Title: Use of Non-invasive Optical Analysis in Neurosurgery - A Pilot Study
Brief Title: Use of Non-invasive Optical Analysis in Neurosurgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 258210
Record Dates: First submitted 2020-03-24; First posted 2021-01-15 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Brain Tumour; Glioma; Meningioma; Brain Metastases; Schwannoma
Keywords: gliomas; multispectral analysis; hyperspectral analysis; fluorescence; brain tumours
MeSH Terms: conditions — Brain Neoplasms; Glioma; Meningioma; Neurilemmoma | interventions — Hyperspectral Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with brain tumours candidate for neurosurgery (Experimental): Patients will be recruited following the inclusion criteria: any patient with a diagnosis of brain tumour, age ranging from 18 with no upper limit, who will agree to the operation and to take part of the present study, will be enrolled. During surgery, multispectral and/or hyper spectral acquisition of images from the surgical field will be performed. Each patient will have an average acquisition of 6 datasets. As each dataset will correspond to an image, this will be divided into many reading regions (from 10 to 20) for a total of approximatively 60 measurements per patient.
  Interventions: Device: Intra-operative multispectral / hyperspectral analysis

INTERVENTIONS:
Device: Intra-operative multispectral / hyperspectral analysis — During surgery, the operating surgeon will be using standard NHS neurosurgical equipment such as an endoscope and/or a microscope. This equipment is operated in exactly the same way as with any other procedure, but either the microscope or the endoscope in use will be connected to the system of camera and filters for multispectral/hyperspectral analysis. During each surgical intervention, tissue-specific spectral data will be collected at specific stages - mostly once the brain surface is exposed and at the end of the resection on the surgical cavity. The operation will be visually recorded in order to sync visual data with the spectral data obtained at the same moment in time. The video recording will not be patient identifiable and will be viewed only by members of the research team working on this project (see below). The use of video recording equipment will be included in the patient information sheet given to all patients prior to gaining consent

SUMMARY:
The present study aims to investigate the potential application of multispectral analysis, hyperspectral imaging, and fluorescence during neuro-oncological procedures, specifically during brain tumour debulking / resection. These optics techniques are entirely non-invasive and consist in camera with a filter to be linked to the standard microsurgical and endoscopic instruments used in theatre. The research procedure consists of images acquisition and data processing, with virtually no additional invasive procedures to be performed on patients.

DETAILED DESCRIPTION:
Surgical resection of brain tumours remains a challenge. While the center of a tumour is easily resectable, its margins are often fading into normal brain, and therefore quite difficult to identify. Moreover, there is now extensive literature proving that tumour cells extend way beyond visible margins of a tumour, following white matter tracts in the brain. As opposite to different organs (such as liver or kidney), resection of brain tumours beyond the visible margins is limited by the presence of eloquent/functional areas. Damages or resection of these areas will inevitably cause a permanent disability, which can be incredibly serious and impact on further treatment: a paralyzed or unconscious patient is not capable of tolerating chemotherapy or radiotherapy after surgery, both crucial complementary forms of treatment to contain the disease, in combination with surgery.

Because of these premises, the concept of "functional margins of resection" is now established in the neurosurgical community: a tumour is resected and the resection is pushed up to 1-2 cms beyond the margins or only up to the point where a functional/eloquent area is found. If the latter is the case, the functional area is obviously preserved and tumour resection is stopped. Identifying these areas is the main challenge in brain tumour surgery.

The aim of this study and its scientific justification is to refine a new, potentially more practical and quick technique to identify functional brain areas in real time. This study can serve as a benchmark study to both improve surgery of brain tumours and increase our knowledge about brain tumours and eloquent brain vascular supply. This technique can also potentially be implemented to obtain a novel technology to assess brain perfusion during neurosurgical procedures. Maintaining blood supply to healthy brain tissue is a key component of successful neuro-oncological surgery. Multispectral/hyperspectral analysis can be evaluated as a complementary tool to assess brain perfusion in real-time and prevent post-operative devastating neurological complications, such as strokes, or significantly reduce the secondary damage would these complications occurr.

The present project consists of a pilot observational study on patients diagnosed with brain tumours candidate for a neurosurgical operation.

From a practical point of view, participation in the study will only imply that some images will be acquired during surgery and processed at a later stage. The study won't impact on patients' care at any stage, nor will produce results that will be relevant for future medical records of patients enrolled. Patients will be approached about this study at the time of their first neuro-oncology clinic consultation. A member of the research team will be present at the time of the consultation and will explain in details what are the purposes and the methods of the present study.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for surgery due to a confirmed clinical and radiological diagnosis of cranial intrinsic or extrinsic tumour - any histological diagnosis confirming neuro-oncological disease, including primary and secondary disease
* Agreed to take part to the present research protocol and signed proper informed consent form

Exclusion Criteria:

* Suspected differential diagnosis of pathological condition affecting central nervous system other than neuro-oncological disease - including demyelinating diseases, infections, brain traumas / haematomas, vascular or auto-immune diseases
* Patients not capable to give consent - not in condition of understanding, processing and retaining information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-28 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Analysis of spectroscopic signal reading between brain tissue and brain tumour | 3 years
  Brain tissue and tumour tissue, the signals collected will be correlated both to the visual signal seen on normal operative field, a pre-set of brain images, and the signal seen on the peri-operative imaging (MRI scan).
Analysis of spectroscopic signal reading between functional brain areas and non functional brain areas | 3 years
  The signal collected will be correlated with the neuro-physiological intra-operative findings, in every case there is an indication to do so, and with the expected location of the eloquent areas on the peri-operative images.

SECONDARY OUTCOMES:
Analysis of spectroscopic signal reading of surgical field as seen at its baseline and under fluorescence-specific light | 3 years
  Comparison will be made between multispectral / hyper spectral acquired images, and the same images acquired with the addition of fluorescence light

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O'Neill, MD, FRCS, Study Chair — Imperial College of London, Charing Cross Hospital
Locations (1):
- Imperial College NHS Trust, Charing Cross Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Behrooz A, Waterman P, Vasquez KO, Meganck J, Peterson JD, Faqir I, Kempner J. Multispectral open-air intraoperative fluorescence imaging. Opt Lett. 2017 Aug 1;42(15):2964-2967. doi: 10.1364/OL.42.002964. PMID 28957220
- [Background] Lu HD, Chen G, Cai J, Roe AW. Intrinsic signal optical imaging of visual brain activity: Tracking of fast cortical dynamics. Neuroimage. 2017 Mar 1;148:160-168. doi: 10.1016/j.neuroimage.2017.01.006. Epub 2017 Jan 4. PMID 28063974
- [Background] Fawzy Y, Lam S, Zeng H. Rapid multispectral endoscopic imaging system for near real-time mapping of the mucosa blood supply in the lung. Biomed Opt Express. 2015 Jul 21;6(8):2980-90. doi: 10.1364/BOE.6.002980. eCollection 2015 Aug 1. PMID 26309761
- [Background] Zhang Y, Wirkert SJ, Iszatt J, Kenngott H, Wagner M, Mayer B, Stock C, Clancy NT, Elson DS, Maier-Hein L. Tissue classification for laparoscopic image understanding based on multispectral texture analysis. J Med Imaging (Bellingham). 2017 Jan;4(1):015001. doi: 10.1117/1.JMI.4.1.015001. Epub 2017 Jan 25. PMID 28149926

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT04712214/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/14/NCT04712214/ICF_001.pdf